CLINICAL TRIAL: NCT02758834
Title: Half-life of Plasma Phytosterols in Very Low-birth-weight Preterm Infants on Routine Parenteral Nutrition With Soy-bean Oil Based Lipid Emulsions
Brief Title: Half-life of Plasma Phytosterols in Preterm Infants on Parenteral Nutrition
Status: Completed | Type: Observational
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Virgilio Paolo Carnielli, MD, Phd, Università Politecnica delle Marche
Other Study IDs: DG-469
Record Dates: First submitted 2016-04-26; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Liver Diseases
Keywords: Preterm Infants; Phytosterols; Parenteral Nutrition
MeSH Terms: conditions — Liver Diseases; Hyperphagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine plasma phytosterols half-lives in preterm infants who received intravenous soy oil-based lipid emulsions.

DETAILED DESCRIPTION:
Several studies reported the relationship between plasma phytosterol concentrations and parenteral nutrition-associated cholestasis (PNAC). Information on plasma phytosterols half-lives in very-low-birth-weight (VLBW) preterm infants on lipid parenteral nutrition (PN) are lacking. In a prospective cohort study, plasma phytosterols (campesterol, stigmasterol and sitosterol) of VLBW preterm infants on routine PN will be measured by gas chromatography-mass spectrometry (GC-MS) during PN administration and after only lipid stopping. Plasma phytosterols half-lives will be calculated from the monoexponential decay curves. Blood samples will be weekly collected from 1st to 7th week of life during routine metabolic tolerance analysis or gas-analysis in order to avoid burden of additional phlebotomy. Samples will be collected in ethylenediaminetetraacetic acid-tubes and immediately centrifugated. Plasma will be stored in pyrogallol added-tubes at -20°C until analysis. Saponification reaction will be done using 5-alpha-cholestane as internal standard.

ELIGIBILITY:
Inclusion Criteria:

* 24 weeks < gestational age < 32 weeks;
* 500 g ≤ birth weight < 1250 g;
* parenteral nutrition with soy oil-based lipid emulsions from the first hours of life;
* parental consent.

Exclusion Criteria:

* length of parenteral nutrition > 24 days;
* severe malformations;
* inborn errors of metabolism;
* severe congenital sepsis;
* liver dysfunctions.

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants (24 weeks < gestational age < 32 weeks; 500 g ≤ birth weight < 1250 g) who received intravenous soy oil-based lipid emulsions from the first hours of life.
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change of plasma phytosterol concentrations in preterm infants during parenteral nutrition and after only lipid stopping. | 7, 14, 21, 28, 35, 42 and 49 days
  Plasma campesterol, stigmasterol and sitosterol concentrations will be measured at 7, 14, 21, 28, 35, 42 and 49 days from PN started. Plasma phytosterol concentrations will be measured by gas chromatography-mass spectrometry. Calibration curves will be used to calculate the phytosterol plasma concentrations (mg/L).

SECONDARY OUTCOMES:
Normal liver function of preterm infants will be define by conjugated bilirubin values from blood samples under 1 mg/dl. | 7 days and 42 days of life
  Eligibility of preterm infants will be related to a normal liver function. Conjugated bilirubin value from blood sample is a good sign of hepatic function. The threshold value was defined to 1 mg/dl. Preterm infants who will have conjugated bilirubin values more of 1 mg/dl will be excluded from the study. The measure of conjugated bilirubin from blood samples will be routinely done at 7 and 42 days of life.
Plasma phytosterols half-lives | After the collection of 3 or more blood samples collected when the lipid infusion is stopped.
  Plasma phytosterol half-lives (days) will be measured using 3 or more plasma phytosterol concentrations calculated after only lipid stopping. Half-life of plasma phytosterols will be calculated from monoexponential decay curves.

CONTACTS AND LOCATIONS:
Overall Officials: Virgilio P. Carnielli, MD, PhD, Principal Investigator — Università Politecnica delle Marche

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nghiem-Rao TH, Tunc I, Mavis AM, Cao Y, Polzin EM, Firary MF, Wang X, Simpson PM, Patel SB. Kinetics of phytosterol metabolism in neonates receiving parenteral nutrition. Pediatr Res. 2015 Aug;78(2):181-9. doi: 10.1038/pr.2015.78. Epub 2015 Apr 21. PMID 25897540
- [Background] Bhattacharyya AK, Connor WE, Lin DS, McMurry MM, Shulman RS. Sluggish sitosterol turnover and hepatic failure to excrete sitosterol into bile cause expansion of body pool of sitosterol in patients with sitosterolemia and xanthomatosis. Arterioscler Thromb. 1991 Sep-Oct;11(5):1287-94. doi: 10.1161/01.atv.11.5.1287. PMID 1911714
- [Background] Lin HJ, Wang C, Salen G, Lam KC, Chan TK. Sitosterol and cholesterol metabolism in a patient with coexisting phytosterolemia and cholestanolemia. Metabolism. 1983 Feb;32(2):126-33. doi: 10.1016/0026-0495(83)90216-0. PMID 6827984
- [Background] Ostlund RE Jr, McGill JB, Zeng CM, Covey DF, Stearns J, Stenson WF, Spilburg CA. Gastrointestinal absorption and plasma kinetics of soy Delta(5)-phytosterols and phytostanols in humans. Am J Physiol Endocrinol Metab. 2002 Apr;282(4):E911-6. doi: 10.1152/ajpendo.00328.2001. PMID 11882512
- [Background] Salen G, Tint GS, Shefer S, Shore V, Nguyen L. Increased sitosterol absorption is offset by rapid elimination to prevent accumulation in heterozygotes with sitosterolemia. Arterioscler Thromb. 1992 May;12(5):563-8. doi: 10.1161/01.atv.12.5.563. PMID 1576118
- [Derived] Pupillo D, Correani A, Biagetti C, D'Ascenzo R, Simonato M, Verlato G, Cogo P, Rocchi MBL, Carnielli VP. Half-life of plasma phytosterols in very low birth weight preterm infants on routine parenteral nutrition with vegetable oil-based lipid emulsions. Clin Nutr. 2018 Feb;37(1):262-269. doi: 10.1016/j.clnu.2016.12.022. Epub 2016 Dec 30. PMID 28063717